CLINICAL TRIAL: NCT03827837
Title: Famitinib Malate Plus Anti-PD1 Therapy (SHR-1210) in Advanced Renal Cell Carcinoma, Urothelial Carcinoma, Advanced Cervical Cancer, Relapse Ovarian Cancer, Endometrial Cancer: Multi-institutional, Open-label, Phase 2 Trial
Brief Title: Famitinib Plus Anti-PD1 Therapy for Advanced Urinary System Tumor, Advanced Gynecological Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-213
Record Dates: First submitted 2018-11-12; First posted 2019-02-04 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Renal Cell Carcinoma; Urothelial Carcinoma; Cervical Cancer; Ovarian Cancer Recurrent; Endometrial Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 combined with Famitinb (Experimental): SHR-1210 + Famitinib
  Interventions: Biological: SHR-1210; Drug: Famitinib

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody
  Other Names: Camrelizumab
Drug: Famitinib — a small-molecule multikinase inhibitor
  Other Names: Famitinib Malate Capsule

SUMMARY:
Phase II multi-chort, adaptive two-stage, open label, nonrandomized study. The aim of our study is to evaluate the efficacy and safety of anti-PD-1 antibody SHR-1210(Camrelizumab) in combination with a small-molecule multikinase inhibitor Famitinib in subjects with advanced RCC/UC/CC/EC and recurrent OC.

chort1: Renal Cell Carcinoma (RCC) chort2: Urothelial Carcinoma(UC) chort3: Ovarian Cancer (OC) chort4: Cervical Cancer (CC) chort5: Endometrial Cancer (EC)

DETAILED DESCRIPTION:
Stage 1: Approximately 110 participants will be recruited, 22 participants per chort; Stage 2: Approximately 55 participants will be recruited, 11 participants per chort, if more than 7（including 7） patients reached ORR in every chort ; Approximately 155 participants will be recruited, 21 participants per chort, if 3 ≤ patients <7 patients reached ORR in every chort.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/ for the trial.
2. Be at least 18 years of age on day of signing informed consent, male or female.
3. Patients with one of the following tumors:

   * Histologically or cytologically confirmed diagnosis of advanced renal cell carcinoma (defined as more than 50% clear cell component) after failure of IL-2 and/or anti-VEGF TKI treatment. If patients didn't want to use anti-VEGF TKI medicine or couldn't stand anti-VEGF TKI medicine costs, they will also be considered.
   * Histologically or cytologically confirmed diagnosis of unresectable urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra (defined as more than 50% transitional cell component) after failure of no more than two prior platinum-based chemotherapeutic regimen.
   * Histologically or cytologically confirmed diagnosis of advanced squamous cell carcinoma of the cervix after failure of first-line system treatment.
   * Histologically confirmed diagnosis of recurrent or refractory epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer that are relapsed and resistant (recurred less than 6 months after chemotherapy) or refractory (progressed on chemotherapy) to prior platinum-based standard care systemic regimen.
   * Histologically confirmed diagnosis of recurrent or refractory endometrial cancer that are relapsed and resistant or refractory (progressed on chemotherapy) to prior platinum-based standard care systemic regimen.
4. At least one measurable lesion according to RECIST 1.1.
5. The patients can swallow pills.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. Life expectancy of at least 12 weeks.
8. The results of patients' blood tests are as follows:-Neutrophils≥1.5E+9/L; - Plt≥90E+9/L; -Hb≥90g/L; -ALB≥30g/L ;-TSH≤1×ULN;-TBIL ≤ 1 ×ULN;-ALT and AST ≤ 3 ×ULN; AKP≤ 2.5×ULN; -Creatinine ≤ 1.5×ULN.
9. Male or Female patient of childbearing potential (entering the study after a menstrual period and who have a negative pregnancy test), who agrees to use two methods (one for the patient and one for the partner) of medically acceptable forms of contraception during the study and for 3 months after the last treatment intake.

Exclusion Criteria:

1. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
2. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
3. Known history of hypersensitivity to other antibody formulation.
4. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 2 weeks prior to trial treatment.
5. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents: systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥ 90 mmHg.
6. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to（1）Congestive heart failure (New York heart association (NYHA) class > 2)；（2）unstable or severe angina; （3）myocardial infarction within 12 months before enrollment；（4） ventricular arrhythmia which need medical intervention.（5）QTc>450ms（male）/QTc>470ms (female)；
7. Coagulation abnormalities (INR>2.0、PT>16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy.
8. Bleeding history, having bleeding event（≥3 Grade according CTCAE 4.0 ）within 4 weeks before screening.
9. Tumor invasion around major vessels shown by imaging, high risk of major vascular invasion leading to massive hemorrhage judged by investigators.
10. Previous Arterial/venous thrombosis events within 6 months.
11. Known hereditary or acquired bleeding and thrombosis tendency.
12. Proteinuria ≥ (++) and 24 hours total urine protein > 1.0 g.
13. Prior chemotherapy, radiotherapy, surgery therapy within 4 weeks or palliative radiotherapy within 2 weeks or target therapy within 5 half-life of the drug before the study drug administration, or any unresolved AEs > Common Terminology Criteria for Adverse Events (CTCAE) Grade 1.
14. Active infection or an unexplained fever > 38.5°C within 7 days before the study drug administration, or baseline WBC>15×E+9/L .
15. Has known history of Interstitial lung disease, or using steroids evidence of active, non-infectious pneumonitis, or would interfere with the detection and handling of suspicious drug-related pulmonary toxicity.
16. History of immunodeficiency or human immunodeficiency virus (HIV) infection.
17. HBV DNA>500 IU/ml，HCV RNA>1000copies/ml，HBsAg+ and anti-HCV+；
18. Has a known additional malignancy within the last 5 years, or that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or patients with recurrent ovarian cancer has a known additional breast cancer that has been radical mastectomy and doesn't relapse within 3 years.
19. Patients with treatment history of SHR-1210 or any other PD-L1 or PD-1 antagonists or famitinib.
20. Patients who may receive live vaccine during the study, or previous had vaccination within 4 weeks.
21. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's safety and participate in the study or would interfere with the interpretation of the results or lead to the trial being terminated early.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  Defined as complete or partial response per RECIST 1.1 criteria with assessment every 9 weeks

SECONDARY OUTCOMES:
Duration of Response (DoR) | Up to 2 years
  Duration of Response (DoR) per RECIST 1.1
Disease Control Rate (DCR) | Up to 2 years
  Disease Control Rate per RECIST 1.1
Time to objective response(TTR) | Up to 2 years
  Time to objective response per RECIST 1.1
Progression-free survival(PFS) | Up to 2 years
  Progression-free survival(PFS) per RECIST 1.1
Overall survival(OS) | Up to 2 years
  Overal Survial will be calculated based on Kaplan-Meier estimates
12-month survival rate | Up to 1 year
  12-month survival rate will be calculated based on Kaplan-Meier estimates of Overall survival at 12 months
number of participants who experience an adverse event (AE) | From the first assignment of informed consent form up to 90 days after the last dose
  number of participants who experience an adverse event (AE) per CTCAE 4.03
serum SHR-1210 concentrations | From the first dose up to 30 days after the last dose
  serum SHR-1210 concentrations
Positive rate of ADA | From the first dose up to 30 days after the last dose
  Positive rate of anti-SHR1210 antibody
Maximum Observed Plasma Concentration (Cmax) | Day 1 of cycle 3 (each cycle is 21 days)
  Cmax, based PK parameters
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day 1 of cycle 3 (each cycle is 21 days)
  Summarized by dose, cycle, day and time
Apparent Oral Clearance (CL/F) | Day 1 of cycle 3 (each cycle is 21 days)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, MD, Principal Investigator — Fudan University; Xiaohua Wu, MD, Principal Investigator — Fudan University
Locations (1):
- Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xia L, Zhou Q, Gao Y, Hu W, Lou G, Sun H, Zhu J, Shu J, Zhou X, Sun R, Wu X. A multicenter phase 2 trial of camrelizumab plus famitinib for women with recurrent or metastatic cervical squamous cell carcinoma. Nat Commun. 2022 Dec 8;13(1):7581. doi: 10.1038/s41467-022-35133-4. PMID 36481736
- [Derived] Qu YY, Sun Z, Han W, Zou Q, Xing N, Luo H, Zhang X, He C, Bian XJ, Cai J, Chen C, Wang Q, Ye DW. Camrelizumab plus famitinib for advanced or metastatic urothelial carcinoma after platinum-based therapy: data from a multicohort phase 2 study. J Immunother Cancer. 2022 May;10(5):e004427. doi: 10.1136/jitc-2021-004427. PMID 35537782
- [Derived] Xia L, Peng J, Lou G, Pan M, Zhou Q, Hu W, Shi H, Wang L, Gao Y, Zhu J, Zhang Y, Sun R, Zhou X, Wang Q, Wu X. Antitumor activity and safety of camrelizumab plus famitinib in patients with platinum-resistant recurrent ovarian cancer: results from an open-label, multicenter phase 2 basket study. J Immunother Cancer. 2022 Jan;10(1):e003831. doi: 10.1136/jitc-2021-003831. PMID 35017154